CLINICAL TRIAL: NCT00991042
Title: Analytical Transversal Study of Cytokines Serum Levels in Chronic Low Back Pain Due to Herniated Disk
Brief Title: Study of Cytokines Serum Levels in Chronic Low Back Pain
Acronym: cytokine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Federal University of Bahia (Other)
Responsible Party: Durval Campos Kraychete, Universidade Federal da Bahia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: cytokine
Record Dates: First submitted 2009-10-06; First posted 2009-10-07 (Estimated); Last update posted 2009-10-07 (Estimated); Status verified 2009-10

CONDITIONS: Interleukines
Keywords: Cytokines; Low back pain; Intervertebral disk displacement; Interleukins; Tumor necrosis factor-alpha
MeSH Terms: conditions — Low Back Pain; Intervertebral Disc Displacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- cytokine levels (Other): Serum levels of pro-inflammatory cytokines were measured using the Enzyme Linked Immuno Sorbent Assay (ELISA) technique in 23 patients with pain due to herniated disk disease (G1) as well as in 10 control healthy subject
  Interventions: Other: blood collect

INTERVENTIONS:
Other: blood collect — Five milliliters of venous blood was drawn in the morning from subjects and immediately centrifuged.
  Other Names: serum levels

SUMMARY:
The purpose of this study is to:

* evaluate if there is an association between elevated levels of cytokines and chronic pain due to herniated disk disease
* measured cytokines levels in chronic low back pain and in healthy subjects.

DETAILED DESCRIPTION:
23 patients with at least three months of back pain due to herniated disk disease were selected Diagnosis was confirmed by magnetic resonance imaging (MRI) or computerized tomography (CT) imaging of the spine for all patients. In addition, pain severity had to be ³ 5 points on the Numerical Rating Scale (NRS) ranging from zero (no pain) to 10 (worst imaginable pain).

The exclusion criteria were defined as one or more of the following: psychiatric disorders, systemic or inflammatory disease, history of allergy, presence of motor deficits, history of blood dyscrasia, pregnancy, active infection, tumor, use of analgesic drugs in the week before or inability to come to the hospital for evaluation.

ELIGIBILITY:
Inclusion Criteria:

* 23 patients

  * least three months of back pain due to herniated disk disease
  * pain severity had to be 5 points on the Numerical Rating Scale (NRS)
* 10 healthy volunteers:

  * without previous history of back pain

Exclusion Criteria:

* One or more of the following:

  * psychiatric disorders
  * systemic or inflammatory disease
  * history of allergy
  * presence of motor deficits
  * history of blood dyscrasia
  * pregnancy
  * active infection, tumor
  * use of analgesic drugs in the week before
  * inability to come to the hospital for evaluation.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2003-08; Primary Completion 2004-09 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
cytokines levels in patients with chronic low back pain and in healthy subjects | 30 days after collect

CONTACTS AND LOCATIONS:
Overall Officials: Durval C Kraychet, Principal Investigator — Federal University of Bahia
Locations (1):
- Universidade Federal da Bahia, Salvador, Estado de Bahia, Brazil